CLINICAL TRIAL: NCT05393245
Title: Safety Profile of Tiotropium + Olodaterol Used as Maintenance Treatment in COPD Patients in Taiwan: a Non-interventional Study Based on the Taiwan National Health Insurance (NHI) Data
Brief Title: Safety of Tiotropium + Olodaterol in Chronic Obstructive Pulmonary Disease (COPD) Patients in Taiwan: a Non-interventional Study Based on the Taiwan National Health Insurance (NHI) Data
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0109
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients treated with tiotropium and olodaterol (Tio+Olo)
  Interventions: Drug: Tiotropium+Olodaterol; Device: Spiolto Respimat
- COPD patients using other Long-acting muscarinic antagonists/Long-acting β2-agonists (LAMA/LABAs)
  Interventions: Drug: Long-acting muscarinic antagonists (LAMAs); Drug: Long-acting β2-agonists (LABAs)

INTERVENTIONS:
Drug: Tiotropium+Olodaterol — Tiotropium+Olodaterol
  Groups: COPD patients treated with tiotropium and olodaterol (Tio+Olo)
Device: Spiolto Respimat — Spiolto Respimat Inhaler device
  Groups: COPD patients treated with tiotropium and olodaterol (Tio+Olo)
Drug: Long-acting muscarinic antagonists (LAMAs) — Long-acting muscarinic antagonists (LAMAs)
  Groups: COPD patients using other Long-acting muscarinic antagonists/Long-acting β2-agonists (LAMA/LABAs)
Drug: Long-acting β2-agonists (LABAs) — Long-acting β2-agonists (LABAs)
  Groups: COPD patients using other Long-acting muscarinic antagonists/Long-acting β2-agonists (LAMA/LABAs)

SUMMARY:
The aim of this real world study is to assess the safety profile of tiotropium/olodaterol (Tio/Olo).

ELIGIBILITY:
Patients treated with Tio+Olo:

Inclusion criteria:

1. At least one prescription for Tio+Olo (fixed dose combination (FDC) or free combination) as a new initiation between 1st January 2014 and 31st December 2019.
2. Aged ≥ 40 years on the index date.
3. At least one diagnosis of COPD at any time prior to or on the index date.
4. At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs.
5. At least one record in the health insurance system database.

Exclusion criteria:

1. Any use of Tio+Olo in free or fixed form within one year prior to the index date.
2. Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date.

Patients using other Long-acting β2-agonists/Long-acting muscarinic antagonists (LAMA/LABAs):

Inclusion criteria:

1. At least one prescription for LAMA+LABA (FDC or free combination) other than Tio/Olo as a new initiation between 1st January 2014 and 31st December 2019.
2. Aged ≥ 40 years on the index date.
3. At least one diagnosis of COPD at any time prior to or on the index date-
4. At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs.
5. At least one record in the health insurance system database.

Exclusion criteria:

1. Any use of LAMA+LABA in free or fixed form for one year prior to the index date.
2. Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with chronic obstructive pulmonary disease (COPD) in routine clinical practice in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 19467 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Data Research Center, National Taiwan University, Taiwan, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study based on existing data from the Taiwan National Health Insurance (NHI) claims data between 2014 and 2019. This study aimed to estimate the incidence of safety outcomes in Chinese patients with chronic obstructive pulmonary disease (COPD) in routine clinical practice in Taiwan who initiated Tiotropium / Olodaterol (Tio/Olo).
Pre-assignment Details: Every patient who fulfilled inclusion and exclusion criteria was selected until the required sample size was achieved.
Groups:
- Tiotropium/Olodaterol (Tio/Olo): Patients with Chronic Obstructive Pulmonary Disease (COPD) new initiators of Tiotropium+Olodaterol (fixed dose combination (FDC) or free combination) between the 1st January 2014 and 31st December 2019 from the Taiwan National Health Insurance (NHI) claims data.
- Other LABA/LAMA: Patients with Chronic Obstructive Pulmonary Disease (COPD) new initiators of other Long-acting β2-agonists + Long-acting muscarinic antagonists (LAMA+LABA) (fixed dose combination (FDC) or free combination) between the 1st January 2014 and 31st December 2019 from the Taiwan National Health Insurance (NHI) claims data.
Period: Overall Study
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Started | 5820 | 13647
Completed | 5820 | 13647
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA | Total
Number analyzed (Participants) | 5820 | 13647 | 19467
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 72 [63 to 82] | 69 [61 to 78] | 70 [62 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 653 | 1384 | 2037
  Male | 5167 | 12263 | 17430
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Adverse Events in Patients With COPD Treated With Tio+Olo: Potentially Recurrent Events
Description: Incidence rate of adverse events in patients with COPD treated with Tiotropium+Olodaterol (Tio+Olo) per number of person-years is reported. From the index date until the earliest: Outcome of interest, disenrollment, the end of the study period, death, discontinuation of the index drug, addition of Inhaled corticosteroids mono on top of Tio/Olo. The incidence rate was reported as (Total number of patients in the Tio+Olo cohort experiencing an event of interest for the 1st time during the given time period) / (Total person-time at risk from current use of Tio+Olo during the given period). Urinary tract infection: (1): Diagnosis codes were primary inpatient diagnosis associated with a hospitalization. (2): Diagnosis codes were primary or secondary diagnosis associated with a hospitalization.(3): Diagnosis codes were primary or secondary diagnosis associated with a hospitalization OR associated with at least 2 outpatient/emergency visits within 30 days of each other.
Time Frame: From index date between 1st January 2014 until 31st December 2019. Up to 2160 days.
Population: Eligible Patients set: All patients who met the criteria and who were treated with Tio/Olo were included in the analysis dataset.
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Tiotropium/Olodaterol (Tio/Olo)
Number analyzed (Participants) | 5820
Events per 100 person-years
  Nasopharyngitis | 10.63 [9.45 to 11.96]
  Pneumonia- Diagnosis codes were primary inpatient diagnosis associated with a hospitalization | 0.55 [0.33 to 0.91]
  Pneumonia-Diagnosis codes were primary or secondary diagnosis associated with a hospitalization | 0.84 [0.56 to 1.26]
  Moderate COPD exacerbation | 19.71 [18.05 to 21.52]
  Severe COPD exacerbation | 15.66 [14.21 to 17.26]
  Constipation | 17.06 [15.53 to 18.74]
  Diarrhoea | 1.58 [1.17 to 2.13]
  Urinary retention | 6.17 [5.30 to 7.19]
  Urinary tract infection (1) | 2.53 [2.00 to 3.21]
  Urinary tract infection (2) | 9.44 [8.34 to 10.68]
  Urinary tract infection (3) | 13.54 [12.20 to 15.03]
  Urticaria | 6.96 [6.02 to 8.04]
  Rash | 0.69 [0.44 to 1.09]

2. Primary Outcome: Incidence Rate of Adverse Events in Patients With COPD Treated With Tio+Olo: Incident Events
Description: Incidence rate of Adverse Events (AEs) in patients with COPD treated with Tiotropium+Olodaterol (Tio+Olo) per number of person-years is reported. From index date until the earliest: Outcome of interest, disenrollment, end of the study period, death, discontinuation, use of Inhaled corticosteroids. Incident events. The incidence rate was reported as (Total number of patients in the Tio+Olo cohort experiencing an event of interest for the 1st time during the given time period) / (Total person-time at risk from current use of Tio+Olo during the given period). Urinary tract infection: (1): Diagnosis codes were primary inpatient diagnosis associated with a hospitalization. (2): Diagnosis codes were primary or secondary diagnosis associated with a hospitalization.(3): Diagnosis codes were primary or secondary diagnosis associated with a hospitalization OR associated with at least 2 outpatient/emergency visits within 30 days of each other.
Time Frame: From index date between 1st January 2014 until 31st December 2019. Up to 2160 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Tiotropium/Olodaterol (Tio/Olo)
Number analyzed (Participants) | 5820
Events per 100 person-years
  Arrhythmia | 6.80 [5.83 to 7.94]
  Myocardial ischemia | 4.02 [3.31 to 4.90]
  Supraventricular tachycardia | 0.33 [0.17 to 0.63]
  Glaucoma | 1.13 [0.79 to 1.62]
  Nonfatal myocardial infarction (1) | 0.59 [0.36 to 0.96]
  Nonfatal myocardial infarction (2) | 1.11 [0.78 to 1.59]
  Nonfatal hemorrhagic stroke (1) | 0.18 [0.08 to 0.44]
  Nonfatal hemorrhagic stroke (2) | 0.66 [0.42 to 1.05]
  Nonfatal ischemic stroke (1) | 1.03 [0.71 to 1.50]
  Nonfatal ischemic stroke (2) | 1.67 [1.25 to 2.24]
  Nonfatal, Acute, but ill-defined, cerebrovascular disease (1) | 0 [0 to 0]
  Nonfatal, Acute, but ill-defined, cerebrovascular disease (2) | 0 [0 to 0]
  Death | 19.15 [17.58 to 20.85]

3. Secondary Outcome: Baseline Characteristics of Patients Who Initiated Tio+Olo or Other LAMA/LABA: Sex
Description: Number of patients by sex according to whether they started Tio+Olo or another LAMA/LABA
Time Frame: At index date between 2014-2019. Up to 2160 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  Male | 5167 | 12263
  Female | 653 | 1384

4. Secondary Outcome: Baseline Characteristics of Patients Who Initiated Tio+Olo or Other LAMA/LABA: Age
Description: Number of patients by age groups according to whether they started Tio+Olo or another LAMA/LABA. The reported age groups are: 40-59, 60-79 and 80+.
Time Frame: At index date between 2014-2019
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  40-59 years old | 905 | 2826
  60-79 years old | 3151 | 8080
  80+ years old | 1764 | 2741

5. Secondary Outcome: Baseline Characteristics of Patients Who Initiated Tio+Olo or Other LAMA/LABA: Calendar Year of Cohort Entry
Description: Number of patients by Calendar year of cohort entry according to whether they started Tio+Olo or another LAMA/LABA. The reported year groups are: 2014, 2015, 2016, 2017, 2018 and 2019.
Time Frame: At index date between 2014-2019
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  2014 | 0 | 218
  2015 | 150 | 945
  2016 | 241 | 2477
  2017 | 908 | 3491
  2018 | 1944 | 3262
  2019 | 2577 | 3254

6. Secondary Outcome: Baseline Characteristics of Patients Who Initiated Tio+Olo or Other LAMA/LABA: Season of Cohort Entry Date
Description: Number of patients by season of cohort entry date according to whether they started Tio+Olo or another LAMA/LABA. The reported seasons are: Spring (Mar-May), Summer (Jun-Aug), Fall (Sep-Nov) and Winter (Dec-Feb).
Time Frame: At index date between 2014-2019
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  Spring | 1535 | 3748
  Summer | 1484 | 3369
  Fall | 1469 | 3273
  Winter | 1332 | 3257

7. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Specific Previous COPD Treatment
Description: Number of patients by specific previous COPD treatment during the 1 year pre-index baseline period according to whether they started Tio+Olo or another LAMA/LABA is reported. The treatments were: Long-acting muscarinic antagonists (LAMA) monotherapy, Long-acting β2-agonists (LABA) monotherapy, Inhaled corticosteroids (ICS) monotherapy, ICS containing therapy and LAMA+LABA free combinations.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  Long-acting muscarinic antagonists (LAMA) monotherapy | 75 | 465
  Long-acting β2-agonists (LABA) monotherapy | 112 | 670
  Inhaled corticolsteroids (ICS) monotherapy | 76 | 44
  ICS containing therapy | 668 | 1318
  LAMA+LABA free combinations | 699 | 0

8. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Use of Other Respiratory Drugs
Description: Number of patients by use of other respiratory drugs during the 1 year pre-index baseline period according to whether they started Tio+Olo or another LAMA/LABA is reported. The treatments were: Mucolytics, Theophylline, Short-acting beta-agonists and Short-acting muscarinic antagonists.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  Mucolytics | 4324 | 9541
  Theophylline | 2468 | 5913
  Short-acting beta-agonists | 1670 | 2719
  Short-acting muscarinic antagonists. | 911 | 1300

9. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Moderate COPD Exacerbation in 1 Year Prior to Index Date
Description: Number of patients by moderate Chronic Obstructive Pulmonary Disease (COPD) exacerbation in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+ according to the frequency of previous acute COPD exacerbation in 1 year for each patient.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 5209 | 12556
  1 | 483 | 968
  2+ | 128 | 123

10. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Severe COPD Exacerbation in 1 Year Prior to Index Date
Description: Number of patients by severe Chronic Obstructive Pulmonary Disease (COPD) exacerbation in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 5222 | 12738
  1 | 520 | 809
  2+ | 78 | 100

11. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: All COPD Exacerbation in 1 Year Prior to Index Date
Description: Number of patients by Chronic Obstructive Pulmonary Disease (COPD) exacerbations in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 4738 | 11791
  1 | 802 | 1548
  2+ | 280 | 308

12. Secondary Outcome: Baseline Period: Characteristics Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Moderate COPD Exacerbation 30 Days Prior to Index Date
Description: Number of patients by moderate Chronic Obstructive Pulmonary Disease (COPD) exacerbation in 30 days prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 30 consecutive days ending the day before the index date. Up to 30 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 5628 | 13115
  1 | 192 | 532
  2+ | 0 | 0

13. Secondary Outcome: Baseline Period: Characteristics Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Severe COPD Exacerbation 30 Days Prior to Index Date
Description: Number of patients by severe Chronic Obstructive Pulmonary Disease (COPD) exacerbation in 30 days prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 30 consecutive days ending the day before the index date. Up to 30 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 5564 | 13111
  1 | 256 | 536
  2+ | 0 | 0

14. Secondary Outcome: Baseline Period: Characteristics Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: All COPD Exacerbation 30 Days Prior to Index Date
Description: Number of patients by Chronic Obstructive Pulmonary Disease (COPD) exacerbations in 30 days prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 30 consecutive days ending the day before the index date. Up to 30 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 5390 | 12612
  1 | 412 | 1002
  2+ | 18 | 33

15. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Hospitalizations Caused by Exacerbation of COPD in 1 Year Prior to Index Date
Description: Number of hospitalizations caused by Chronic Obstructive Pulmonary Disease (COPD) exacerbations in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 5475 | 13149
  1 | 296 | 443
  2+ | 49 | 55

16. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: All-cause Hospitalizations in 1 Year Prior to Index Date
Description: Number of all-cause hospitalizations in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. Categorized as 0, 1, or 2+.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  0 | 3405 | 9273
  1 | 1311 | 2902
  2+ | 1104 | 1472

17. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Comorbidities in 1 Year Prior to Index Date
Description: Number of participants with comorbidities in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. The following comorbidities are reported: Cardiovascular disease, Cerebrovascular disease, Diabetes, Chronic kidney disease, Pneumonia, Cancer and Cirrhosis.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  Carrdiovascular disease | 2979 | 5741
  Cerebrovascular disease | 857 | 1155
  Diabetes | 1217 | 2407
  Chronic kidney disease | 58 | 224
  Pneumonia | 71 | 218
  Cancer | 274 | 469
  Cirrhosis. | 119 | 279

18. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: Charlson Comorbidity Index (CCI) in 1 Year Prior to Index Date
Description: Charlson Comorbidity Index (CCI) according to whether they started Tio+Olo or another LAMA/LABA is reported.
  The CCI (using Deyo version) is a comorbidity index used to evaluate survival rate in patients with multiple comorbidities. 17 comorbidities were assessed with different weights, and the total score was determined by adding the scores of each comorbidity. The total score goes from 0 to 37, with higher values predicting a higher mortality rate.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Score on a scale | 1.33 (1.14) | 0.97 (1.02)

19. Secondary Outcome: Baseline Period: Characteristics 1 Year Pre-index Comparison Between Patients Who Initiated Tio+Olo or Other LAMA/LABA: History of Medications Dispensed in 1 Year Prior to Index Date
Description: Number of participants with history of medications dispensed in 1 year prior to index date according to whether they started Tio+Olo or another LAMA/LABA is reported. The following medications are reported: Antihypertensives, Antiarrhythmics, Nitrates, Heart failure medications, Lipid-lowering medications, Blood glucose-lowering medications, Anticoagulants and antiplatelet agents, Antibiotics and Antineoplastic agents.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date. Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium/Olodaterol (Tio/Olo) | Other LABA/LAMA
Number analyzed (Participants) | 5820 | 13647
Participants
  Antihypertensives | 4027 | 8720
  Antiarrhythmics | 2192 | 2192
  Nitrates | 1064 | 2227
  Heart failure medications | 2004 | 4086
  Lipid-lowering medications | 1636 | 3823
  Blood glucose-lowering medications | 1386 | 2785
  Anticoagulants and antiplatelet agents | 2473 | 5073
  Antibiotics | 4127 | 9103
  Antineoplastic agents. | 286 | 502

ADVERSE EVENTS:
Time Frame: From index date between 1st January 2014 until 31st December 2019. Up to 2160 days.
Description: The primary objective of the study was to explore the safety outcomes of Tiotropium/Olodaterol, so safety information was extracted from existing data only on these patients. Adverse Events (AEs) on patients treated with Other LABA/LAMA was not collected, only baseline characteristics were collected on these patients. Only AEs pre-specified in the protocol and deaths are reported. Seriousness of AEs was not collected. All patients who met the criteria were included in the analysis dataset
Arm/Group | Tiotropium/Olodaterol (Tio/Olo)
All-Cause Mortality (participants affected / at risk) | 526/5820
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 2014/5820
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium/Olodaterol (Tio/Olo) (N=5820)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 904
Constipation (Gastrointestinal disorders) | 435
Urinary tract infection (Infections and infestations) | 675

LIMITATIONS AND CAVEATS:
According to Boehringer Ingelheim's internal policy, no document date is required in the title page of the Statistical and Epidemiological Analysis Plan.

A direct comparison of the incidence of AEs in similar studies should take into account that the cohorts in the current study were not matched, and, as a consequence, patients treated with Tiotropium/Olodaterol or Other LABA/LAMA presented different baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT05393245/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT05393245/SAP_001.pdf